CLINICAL TRIAL: NCT00474032
Title: Efficacy of Botox in Patients With Idiopathic Clubfoot
Brief Title: Using Botox to Treat Patients With Idiopathic Clubfoot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H01-70210
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Clubfoot
Keywords: Idiopathic clubfoot; Botox injection; Idiopathic Talipes Equinovarus, also known as Idiopathic clubfoot
MeSH Terms: conditions — Clubfoot | interventions — Botulinum Toxins; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Botulinum Toxin (Type A) injection (10 U/Kg) — See Detailed Description.

SUMMARY:
The purpose of this study is to determine the effectiveness of treatment of idiopathic clubfoot utilizing Botulinum Toxin Type A (Botox). This is not a hypothesis-generating study as we are reporting on outcomes of patients who have been treated by this method of clubfoot treatment.

DETAILED DESCRIPTION:
Subjects with clubfoot will be assessed at the initial visit by Dr. Alvarez. During this visit, the first part of treatment, which is manipulation and casting of the clubfoot will be started. Following this visit, there will be weekly visits for continued manipulation and casting until no further correction of the clubfoot is seen. At this point, (usually after four weeks of casting or when the subject is 6-8 weeks of age), Botox® will be injected into the calf muscles of the affected foot or feet. Before the injection, the patch of skin overlying the intended site(s) of injection will be covered with a local anaesthetic cream (EMLA). This will be applied 30 minutes prior to the injection. This helps numb the skin where the injection will take place. A dose of 10 IU/kg Botox® will be used.

Following the Botox injection another cast will be applied. This will be followed by at least 3 more weekly cast changes to maintain the correction. After the casting and once the child's foot (feet) are big enough and have achieved a minimum of 15 degrees of ankle dorsiflexion with the knee in flexion, the bracing period will begin. This involves use of boots and bars which are worn fulltime until the child begins to weight-bear (usually occurs between 4 to 6 months of age). Until the child reaches skeletal maturity, there will always be a tendency for the foot to return to its clubbed position. Therefore, continued vigilance is part of the care for clubfoot. The following is the appointment schedule, assuming that there are no recurrences:

* Weekly appointments for 3 - 5 weeks for initial manipulation and casting
* Botox® injection
* Weekly appointments for 3 - 4 weeks for casting post Botox® injection or until the foot is big enough to fit in the brace
* Weekly appointments for 10 weeks (brace wear at this point)
* Monthly appointments for 9 months (brace wear at this point)
* Appointments every 6 months until your child reaches 8 years of age
* Yearly appointments thereafter until your child reaches 14 years or skeletal maturity

If there is a recurrence of clubfoot malposition, manipulation and casting will be reinstated and a possible repeat of injection of Botox® will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic clubfoot or clubfoot that is not associated with any other neuromuscular disorders or syndromes

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2003-03; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Surgery rate at any point

SECONDARY OUTCOMES:
Range of motion of treated feet at any follow up

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada